CLINICAL TRIAL: NCT01618058
Title: A Long-Term Observational Cohort Study of HIV Infection in Participants Who Seroconvert After Enrolment in Dapivirine Vaginal Ring Trials
Brief Title: Observational Study of HIV Infection in Participants of Seroconvert During Dapivirine Vaginal Ring Trials
Status: Completed | Type: Observational
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IPM 007
Record Dates: First submitted 2012-06-08; First posted 2012-06-13 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: HIV Infections
Keywords: HIV Infections; Anti-HIV Agents; HIV-1
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ARV-Treated Participants: Those participants who received dapivirine during HIV seroconversion
  Interventions: Drug: No Investigational Product
- ARV-Naive Participants: Those participants who received placebo during HIV seroconversion
  Interventions: Drug: No Investigational Product

INTERVENTIONS:
Drug: No Investigational Product — This study is observational in nature and no investigational product will be used.
  Groups: ARV-Treated Participants, ARV-Naive Participants

SUMMARY:
The purpose of this trial is to determine if exposure to ARV-containing investigational products in IPM clinical trials will impact the natural history of HIV infection as measured by the virologic, immunologic and clinical outcomes of participants who become HIV-positive during the IPM 027 trial.

ELIGIBILITY:
Inclusion Criteria:

* Recent HIV seroconversion during participation in IPM 027, according to the HIV testing algorithm of that trial
* Ability and willingness to provide informed consent
* Willingness to give the research centre permission to share information with the primary health care provider (PHCP), and willingness to sign approved site-specific documentation to facilitate such sharing.

Exclusion Criteria:

* Any condition that, in the opinion of the Investigator, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Both microbicide and placebo recipients in IPM 027 who have become HIV infected (HIV-1 or HIV-2) while participating in IPM 027 will be offered enrolment in IPM 007 at the exit visit of IPM 027, i.e. approximately 6 weeks after identification of HIV seroconversion.
  This study includes all active IPM clinical research centres that enrol participants for IPM microbicide trials.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2012-10-04 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
To identify HIV drug resistant mutations following recent seroconversion in plasma and vaginal secretions and change in resistant mutations over time in participants previously exposed to an ARV-based microbicide or a placebo. | 12 months
  The primary outcome will be assessed by viral genotype assay at baseline and at exit from the protocol, to assess the occurrence and frequency of acquiring a drug resistant HIV virus during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Linda-Gail Bekker, Study Chair — Desmond Tutu HIV Centre
Locations (5):
- Project Ubuzima, Kiyovu, Kigali, Rwanda
- South Africa (4):
  - Qhakaza Mbokodo, Ladysmith, KwaZulu-Natal
  - Prevention for HIV and AIDS Project (PHIVA), Pinetown, KwaZulu-Natal
  - Madibeng Centre for Research (MCR), Brits
  - Maternal, Adolescent and Child Health (MatCH), Plessislaer

REFERENCES:
- [Derived] Steytler J, van der Ryst E, Craig C, Van Baelen B, Nuttall J, van Niekerk N, Mellors J, Parikh U, Wallis C; IPM 007 Study Team. Clinical Presentation, Treatment Response, and Virology Outcomes of Women Who Seroconverted in the Dapivirine Vaginal Ring Trials-The Ring Study and DREAM. Clin Infect Dis. 2023 Feb 8;76(3):389-397. doi: 10.1093/cid/ciac804. PMID 36189636